CLINICAL TRIAL: NCT00406068
Title: Open-label, Multi-center Study of the Efficacy and Safety of MCC in the Treatment of Patients With Non-muscle Invasive (Superficial) Bladder Cancer at High Risk of Progression and Who Are Refractory to BCG
Brief Title: Mycobacterial Cell Wall-DNA Complex in Treatment of BCG-refractory Patients With Non-muscle Invasive Bladder Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bioniche Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIS-0611-0602
Record Dates: First submitted 2006-12-01; First posted 2006-12-04 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Bladder Neoplasms
Keywords: Bladder neoplasm; Intravesical drug administration; Neoplasm recurrence, local; Transitional cell, carcinoma; Carcinoma in situ; Mycobacterium
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasm Recurrence, Local; Carcinoma, Transitional Cell; Carcinoma in Situ; Mycobacterium Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mycobacterial cell wall-DNA complex (Experimental): Mycobacterial cell wall-DNA complex
  Interventions: Drug: Mycobacterial cell wall-DNA complex

INTERVENTIONS:
Drug: Mycobacterial cell wall-DNA complex — 8 mg MCC, intravesical - Induction Phase (6 weekly intravesical instillations) and Maintenance Phase (3 weekly instillations at months 3, 6, 12, 18 and 24).
  Other Names: MCC - Urocidin

SUMMARY:
The purpose of this study is to determine the efficacy and safety of intravesical Mycobacterial Cell Wall-DNA Complex (MCC) in patients with non-muscle invasive transitional cell carcinoma (papillary tumors and/or carcinoma in situ) of the urinary bladder at high risk of progression who are refractory to therapy with bacillus Calmette-Guerin (BCG).

DETAILED DESCRIPTION:
The study will be divided into 3 phases: Induction, Maintenance, and Follow-up.

The Induction Phase will cover a period of 6 weeks. During this time, patients will receive 6 weekly intravesical instillations of 8 mg MCC. The patients will be evaluated at month 3, at which time the patients will enter the Maintenance Phase. The Maintenance Phase will last from month 3 to month 24, and during this time, patients will receive weekly MCC instillations for three weeks at months 3, 6, 12, 18, and 24 and evaluations will be performed at months 3, 6, 9, 12, 15, 18, 21 and 24.

At month 3, the patient will be evaluated to assure that the disease is not progressing. Cytology, cystoscopy and biopsies will be performed to obtain adequate staging (if residual tumor persists). If the patient is disease-free, maintenance therapy will be initiated. Patients with non-muscle invasive tumors at month 3 will, at the discretion of the investigator, receive either a second 6-week induction course or a 3-week maintenance course. Patients who show progression to muscle invasive disease will be referred to other treatments.

At month 6 and thereafter at each evaluation visit, patients will be evaluated and managed according to the following results:

* Patients who are disease-free will continue on maintenance treatment.
* Patients who are not disease-free (evidence of papillary lesions, CIS or muscle invasive disease) will be withdrawn from further study treatment and will be referred to other therapies at the discretion of the investigator.

The final 36 months of the study is the Follow-up Phase. Evaluations will be performed at months 30, 36, 42, 48, 54 and 60.

Efficacy evaluations will include standard cystoscopy, biopsies and urine cytology. During the Maintenance Phase, standard cystoscopies will be performed at months 3, 6, 9, 12, 15, 18, 21 and 24 for the surveillance of bladder tumors. During the months that instillations will be performed, cystoscopies will be conducted only once at each of these months. During the Follow-up Phase, cystoscopies will be performed at months 30, 36, 42, 48, 54 and 60.

Mandatory bladder biopsies will be done for all patients at month 6.

During the course of the study, biopsies will be taken only if evident or suspicious lesions are seen during cystoscopy or in case of negative cystoscopy but positive cytology.

ELIGIBILITY:
Inclusion Criteria:

* Patients refractory to BCG therapy;
* Patients with histologically confirmed diagnosis of high grade lesions;
* Diagnosis of high grade lesion must be within 56 days prior to beginning of study treatment;
* Have had all visible papillary lesion(s) resected by TURBT within 56 days prior to beginning of study treatment;
* Available for the whole duration of the study including follow-up (60 months);
* Life expectancy of > 5 years;
* Patients with an ECOG performance status grade of 2 or less;
* Absence of urothelial carcinoma involving the upper urinary tract or prostatic urethra within 12 months from beginning of study treatment;
* Able to understand and give written informed consent;
* In the investigator's judgment, the patient is able to participate in the study.

Exclusion Criteria:

* Current or previous history of muscle invasive tumors;
* Current or previous history of lymph node or distant metastases from bladder cancer;
* Current systemic cancer therapy;
* Current or prior pelvic external beam radiotherapy;
* Pelvic brachytherapy within 2 years of study entry;
* Prior treatment with MCC;
* Patients with existing urinary tract infection or recurrent severe bacterial cystitis;
* Clinically significant and unexplained elevations of liver or renal function tests;
* White blood cell count below 3 x109/L (3,000/mm3) or platelet count below 100 x 109/L(100,000/mm3);
* Severe cardiovascular disease;
* Women who are pregnant or lactating;
* Congenital or acquired immune deficiency;
* With history of malignancy of any organ system, treated or untreated, within the past 5 years (with the exception of adequately treated basal cell or squamous cell carcinoma of the skin, stage T1 prostate cancer, carcinoma in situ of the cervix or colon polyps);
* Previous investigational treatment within 3 months from beginning of study treatment;
* Patients who cannot hold the instillation for one hour;
* Patients who cannot tolerate intravesical administration or intravesical surgical manipulation (cystoscopy or biopsy);
* Clinically significant active infections;
* Any medical or psychiatric condition which, in the opinion of the investigator, would preclude the participant from adhering to the protocol or completing the trial per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2006-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
One year disease-free survival rate | Prospective

SECONDARY OUTCOMES:
The 3, 6 and 24 month disease-free survival rate | Prospective
Duration of disease-free survival in all patients | Prospective
Time to progression to muscle invasive disease | Prospective
Overall survival in all patients | Prospective
Rate of overall drug-related adverse events leading to two consecutive treatment delays of one week each or to the discontinuation of treatment. | Prospective

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Morales, MD, Principal Investigator — Centre for Applied Urological Research, Kingston General Hospital/Queen's University
Locations (31):
- United States (20):
  - BCG Oncology, Phoenix, Arizona
  - San Diego Clinical Trials, San Diego, California
  - Connecticut Urological Research at Grove Hill, New Britain, Connecticut
  - University of Miami School of Medicine, Miami, Florida
  - Winter Park Urology Associates P.A., Orlando, Florida
  - The University of Chicago Hospitals, Chicago, Illinois
  - Welborn Clinic, Evansville, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Chesapeake Urology Research Associates, Towson, Maryland
  - Sheldon J Freedman, MD, Ltd, Las Vegas, Nevada
  - Delaware Valley Urology, LLC-Voorhees, Voorhees Township, New Jersey
  - Memorial Sloan Kettering Cancer Centre, New York, New York
  - Hudson Valley Urology, Poughkeepsie, New York
  - University of Rochester Medical Center, Rochester, New York
  - Triangle Urology Group, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Urology Clinics of North Texas, P.A., Dallas, Texas
  - M.D. Anderson Cancer Center, Houston, Texas
  - Urology San Antonio Research, PA, San Antonio, Texas
  - Sentara Medical Group - Urology of Virginia, PC, Norfolk, Virginia
- Canada (11):
  - Andreou Research, Surrey, British Columbia
  - Can-Med Clinical Research, Victoria, British Columbia
  - Dr. Steinhoff Clinical Research, Victoria, British Columbia
  - Centre for Applied Urological Research, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network / Princess Margaret Hospital, Toronto, Ontario
  - The Male Health Center, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Centre de Recherche du CHUQ, Québec, Quebec

REFERENCES:
- [Result] Morales A, Herr H, Steinberg G, Given R, Cohen Z, Amrhein J, Kamat AM. Efficacy and safety of MCNA in patients with nonmuscle invasive bladder cancer at high risk for recurrence and progression after failed treatment with bacillus Calmette-Guerin. J Urol. 2015 Apr;193(4):1135-43. doi: 10.1016/j.juro.2014.09.109. Epub 2014 Oct 5. PMID 25286009